CLINICAL TRIAL: NCT01571869
Title: Influence of a Meal on the Efficacy of Plant Sterol Given at Different Times of the Day in Management of Hypercholesterolemia
Brief Title: Pilot Study in the Cholesterol Absorption Reduction After Consumption of Low-fat, Drinkable Fermented Milk Enriched With Plant Sterols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: NU142
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Mildly Hypercholesterolemic Subjects
Keywords: Plant sterol - hypercholesterolemia - dairy - meal
MeSH Terms: interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Experimental)
  Interventions: Other: 1- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) per unit
- 2 = Control product (Placebo Comparator)
  Interventions: Other: 2- Low fat drinkable fermented dairy product without plant sterols (control)

INTERVENTIONS:
Other: 1- Low fat drinkable fermented dairy product enriched with 1.6g of plant sterol (as free equivalent) per unit — 1-Intervention with test product (morning, evening or snack)
  Arms: 1 = Tested product
Other: 2- Low fat drinkable fermented dairy product without plant sterols (control) — 2 - Intervention with control product (morning and/or evening)
  Arms: 2 = Control product

SUMMARY:
The objective of this study is to compare efficacy of a plant sterol enriched yogurt given at different moments of the day in lowering blood cholesterol of hypercholesterolemic.

ELIGIBILITY:
Inclusion Criteria:

* male and post-menopausal female aged 40-80 years;
* BMI between 22 and 32 kg/m2,
* Non-smoker, Stabilized LDL-c over 3.0 mmol/L,
* Not taking any medication known to affect lipid metabolism for at least the previous 3 month period,
* Agree to follow the dietary recommendations in the context of their hypercholesterolemia,
* Have to give written consent to take part in the study

Exclusion Criteria:

* Thyroid disease, diabetes mellitus, kidney disease or liver disease, Hypertension (95<SBP>140 mmHg and/or 45<DBP>90 mmHg),
* Previous history of symptomatic vascular disease, TG level > 2,8 g/l,
* History of metabolic or gastrointestinal disease with the exception of appendicectomy,
* Consumption of large amounts of alcohol,
* Having undergone general anesthesia in the month prior to pre-selection,
* Receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters,
* Having serious or acute disease likely to influence study results or involved in life time,
* Presenting allergy or hypersensitivity to milk proteins, or refusing to consume them,
* Refusing to stop his/her consumption of enriched plant sterol trade products during the study,
* In a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject,
* For female subjects: likely to change her hormonal substitutive treatment,
* Currently in an exclusion period following participation in another clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2005-12 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Ste-anne-de-bellevue, Quebec, Canada